CLINICAL TRIAL: NCT01031095
Title: A RandomisED StUdy Comparing Standard Systemic Anticoagulation ThErapy to Low Dose Intracoronary Anticoagulation Therapy for Elective Percutaneous Coronary Intervention
Brief Title: (A Novel Pharmacologic Regime for Elective Percutaneous Coronary Intervention)
Acronym: REDUCED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Bursa Postgraduate Hospital, Bursa Postgraduate Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BYİEAH1
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; low dose intracoronary heparin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose intracoronary heparin (Experimental): Low dose intracoronary heparin: In this group elective coronary intervention was performed with low dose intracoronary Heparin
  Interventions: Other: coronary intervention
- Standard treatment arm (Active Comparator): Standard treatment arm: In this group elective coronary intervention performed with standard dose intravenous heparin
  Interventions: Other: coronary intervention

INTERVENTIONS:
Other: coronary intervention — elective coronary intervention

SUMMARY:
The hypothesis:

Low dose intracoronary unfractionated heparin is as effective and safe as standard dose intravenous unfractionated heparin on patients with elective percutaneous coronary intervention.

DETAILED DESCRIPTION:
Aim:

Primary objective:To evaluate the efficiency and safety of low dose intracoronary unfractioned heparin (UFH) on elective percutaneous coronary intervention (PCI).

Secondary objective:

* To evaluate the effect of low dose intracoronary UFH on myocardial ischemia after PCI.
* To evaluate the effect of low dose intracoronary UFH on bleeding complications after PCI.
* To evaluate the cost-effectivity of low dose intracoronary UFH on elective PCI

Study central:

* Bursa Postgraduate Hospital, Cardiology Clinic

Study population:

* we planned to enrol 200 patients.
* Patients will randomise in two groups (control group:100 patients, study group:100 patients)

Study works:-Write case report form for all patients

* Control for inclusion criteria
* Demographic data (age, gender)
* Height, weight, BMI and glomerular filtration rate (GFR)
* Risk factors
* laboratory data (biochemical and hematologic)
* Medication history
* Echocardiographic data
* Angiographic data
* Procedure time
* PCI data(vessel diameter, stent diameter, lesion and stent length, performed percutaneous transluminal coronary angioplasty (PTCA) or not, etc)
* Before and after procedure (activated clotting time) ACT value
* Before and after procedure troponin I (TnI) and Creatine kinase MB (CKMB) levels
* Note complication (MACE, bleeding, hematoma etc)
* Note femoral compression time.

  4 weeks later note the first control data.

Six months later note the second control data.

ELIGIBILITY:
Inclusion Criteria:

* The patients; who have planned elective PCI and have had written informed consent for participation to study.
* The native coronary artery;

  * lesion with narrowing >=70%,
  * lesion without thrombus
  * no left main coronary artery (LMCA) lesion
  * no chronic total occlusion lesion

Exclusion Criteria:

* Patients have allergy for acetylsalicylic acid (ASA), Clopidogrel and heparin
* Patients who performed primary PCI
* Patients with acute coronary syndrome
* Patients with have a history of myocardial infarction (MI) for two weeks
* Patients who were use UFH or low molecular weight heparin (LMWH) for 24 hours
* Patients on warfarin therapy
* Patients who have bleeding diathesis, or have high risk for bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Arı, MD, Study Director — Bursa Postgraduate Hospital
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Stabile E, Nammas W, Salemme L, Sorropago G, Cioppa A, Tesorio T, Ambrosini V, Campopiano E, Popusoi G, Biondi Zoccai G, Rubino P. The CIAO (Coronary Interventions Antiplatelet-based Only) Study: a randomized study comparing standard anticoagulation regimen to absence of anticoagulation for elective percutaneous coronary intervention. J Am Coll Cardiol. 2008 Oct 14;52(16):1293-8. doi: 10.1016/j.jacc.2008.07.026. PMID 18929239
- [Derived] Ari H, Kivac E, Ari S, Emlek N, Cetinkaya S, Celiloglu N, Sarigul OY, Aydin C, Akkaya M, Koca V, Bozat T, Gurdogan M. The REDUCED (a RandomisED stUdy Comparing standard systemic anticoagulation thErapy to low Dose intracoronary anticoagulation therapy for elective percutaneous coronary intervention) trial. A novel pharmacologic regime for elective percutaneous coronary intervention. Acta Cardiol. 2014 Dec;69(6):619-27. doi: 10.1080/ac.69.6.1000004. PMID 25643432

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Intracoronary Heparin: Low dose intracoronary heparin treatment arm
- Standard Therapy: standard unfractionated heparin (UFH) treatment
Period: Overall Study
Arm/Group | Low Dose Intracoronary Heparin | Standard Therapy
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Therapy: standard UFH treatment
- Total: Total of all reporting groups
Arm/Group | Low Dose Intracoronary Heparin | Standard Therapy | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 80 | 160
  >=65 years | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.11 (9.68) | 58.99 (11.24) | 59.06 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 75 | 81 | 156
Region of Enrollment [Number; unit: participants]
  Turkey | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac Events
Time Frame: 30 days
Measure: Number; unit: percentage of event
Groups:
- Standard Therapy: standard UFH treatment (intravenous standard dose unfractioned heparin group)
Arm/Group | Standard Therapy
Number analyzed (Participants) | 100
percentage of event | 2

2. Primary Outcome: Major Adverse Cardiac Event
Time Frame: 30 days
Measure: Number; unit: percentage of event
Groups:
- Low Dose Intracoronary Heparin Treatment Arm: low dose intracoronary heparin treatment arm (intracoronary 1000 IU unfractioned heparin arm)
Arm/Group | Low Dose Intracoronary Heparin Treatment Arm
Number analyzed (Participants) | 100
percentage of event | 1

ADVERSE EVENTS:
Arm/Group | Low Dose Intracoronary Heparin | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 1/100 | 2/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Intracoronary Heparin (N=100) | Standard Therapy (N=100)
MI (Cardiac disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The intraprocedural use of a heparinised flush was not controlled; however, given the maximum amount that was allowed to be used, this is not likely to have significantly affected the activated clotting times. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No